CLINICAL TRIAL: NCT05329532
Title: A Phase 1/2, Multicentre, Open-Label Study of Modi-1 Moditope in Patients With Breast, Head and Neck, Ovarian, or Renal Cancer
Brief Title: Modi-1 Moditope in Breast, Head and Neck, Ovarian, or Renal Cancer
Acronym: ModiFY
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Scancell Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Modi-1-001
Record Dates: First submitted 2022-01-31; First posted 2022-04-15 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Triple Negative Breast Cancer; Renal Cell Cancer; High Grade Ovarian Serous Adenocarcinoma; Squamous Cell Carcinoma of the Head and Neck
Keywords: vaccine; peptide; Phase II
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Carcinoma, Renal Cell; Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Open label, uncontrolled study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Patients with TNBC, advanced/unresectable SCCHN, high grade serous ovarian carcinoma, or RCC (Experimental): Modi-1 Moditope Monotherapy
  Interventions: Biological: Modi-1 Moditope; Device: MicronJet600™ microneedle device (NanoPass)
- Patients with advanced/unresectable SCCHN or RCC eligible for standard of care checkpoint inhibitors (Experimental): Modi-1 Moditope + Standard of Care Checkpoint Inhibitors
  Interventions: Biological: Modi-1 Moditope; Device: MicronJet600™ microneedle device (NanoPass)
- Patients with SCCHN eligible for curative intent resection surgery (neoadjuvant cohort) (Experimental): Modi-1 Monotherapy vs Modi-1 Moditope + Pembrolizumab
  Interventions: Biological: Modi-1 Moditope; Biological: Pembrolizumab; Device: MicronJet600™ microneedle device (NanoPass)

INTERVENTIONS:
Biological: Modi-1 Moditope — Modi-1 Moditope administered intradermally (i.d.) using the MicronJet600™ microneedle device (NanoPass).
Biological: Pembrolizumab — Pembrolizumab (exploratory cohorts) will be administered by intravenous infusion on Day 8, prior to tumour resection surgery at 6 weeks.
  Arms: Patients with SCCHN eligible for curative intent resection surgery (neoadjuvant cohort)
Device: MicronJet600™ microneedle device (NanoPass) — Intradermal injection device

SUMMARY:
The main objectives of this study are to assess the safety, tolerability, immunological activity, and preliminary efficacy of the Modi-1 Moditope vaccine, both as monotherapy and in combination with a checkpoint inhibitor (CPI) such as pembrolizumab or nivolumab with or without Ipilimumab (where these are standard of care in a non-neoadjuvant setting), in patients with advanced triple negative breast cancer (TNBC), advanced/unresectable human papillomavirus-negative squamous cell carcinoma of the head and neck (SCCHN), high grade serous ovarian carcinoma (HGSOC), or renal cell carcinoma (RCC).

Modi-1 Moditope will also be investigated in the neoadjuvant setting for patients with SCCHN undergoing curative intent surgical resection in combination with pembrolizumab versus the Modi-1 alone.

DETAILED DESCRIPTION:
This is an open-label, parallel arm, Phase 1/2 study to assess the safety, tolerability, immunological activity, and preliminary efficacy of the Modi-1 Moditope vaccine in patients with advanced TNBC, advanced/unresectable SCCHN, HGSOC, or RCC.

Modi-1 Moditope vaccines, consist of a combination of specific peptides conjugated to a toll-like receptor ligand 1/2 adjuvant, designed to enhance immune responses against peptides commonly expressed or upregulated by cancer cells. Thus, improving immune recognition of these cancers and potentially increasing response rates in patients with advanced solid tumours.

The aim of this study is to investigate preliminary efficacy of Modi-1 Moditope, in an open labelled clinical trial, in participants with TNBC, SCCHN, RCC and HGSOC, powered to demonstrate that Modi-1 Moditope have potent anti-tumour activity.

In this trial, Modi-1 Moditope will be administered, either as monotherapy or in combination with a CPI (as standard of care).

In addition, an exploratory, randomised cohort will be included to assess the impact of Modi-1 Moditope (with or without pembrolizumab) in participants with SCCHN scheduled for resection surgery with curative intent.

Modi-1 Moditope will be administered intradermally using the MicronJet600™ microneedle device referred to as NanoPass.

The study aims to enrol 168 (138 in non-neoadjuvant cohorts and 30 in the exploratory neoadjuvant SCCHN cohort) individuals across multiple UK collaborating clinical centres.

ELIGIBILITY:
INCLUSION CRITERIA

1. Patient either has one of the following histologically or cytologically confirmed advanced cancers not amenable to curative intent surgical resection:

   * TNBC
   * SCCHN (oral cavity, oropharynx, hypopharynx, or larynx)
   * HGSOC including fallopian tube and primary peritoneal cancers
   * RCC Or the patient has histologically or cytologically confirmed SCCHN scheduled to have curative intent surgical resection.
2. Patient must meet one of the following specific criteria for prior treatment of the relevant tumour type:

   * TNBC:

     * patient has received available standard therapy for advanced disease (Modi-1ev/Modi-1eKv monotherapy cohort only).
     * patient stopped immunotherapy due to toxicity and with residual disease as measurable by RECIST 1.1 (Modi-1ev/Modi-1eKv monotherapy cohort only).
     * patient completing a systemic treatment regimen with immunotherapy, for whom a subsequent SOC therapy is not yet indicated or appropriate and with measurable disease in accordance with RECIST 1.1 (Modi-1ev/Modi-1eKv monotherapy cohort only).
     * patient has refused SOC therapy (Modi-1ev/Modi-1eKv monotherapy cohort only).
   * SCCHN:

     * patient has received first-line platinum-containing chemotherapy (with or without radiotherapy) as treatment for advanced disease (Modi-1ev/Modi-1eKv monotherapy and Modi-1ev/Modi-1eKv + CPI cohorts).
     * patient with locally advanced or metastatic disease measurable by RECIST 1.1 for whom all forms of platinum-based chemoradiotherapy treatment are contraindicated (Modi-1ev/Modi-1eKv monotherapy and Modi-1ev/Modi-1eKv + CPI cohorts).
     * patient completing immunotherapy for whom a subsequent SOC therapy is not yet indicated or appropriate and with measurable disease in accordance with RECIST 1.1 (Modi-1ev/Modi-1eKv monotherapy cohort only).
     * patient stopped immunotherapy due to toxicity or completion of immunotherapy but with measurable disease in accordance with RECIST 1.1 (Modi-1ev/Modi-1eKv monotherapy cohort only).
     * patient with untreated metastatic or unresectable recurrent SCCHN whose tumours express PD-L1 with a combined positive score (CPS) of one or more and are eligible for SOC immunotherapy (Modi-1ev/Modi-1eKv + CPI cohort only). Patients who received their first dose of CPI therapy within 28 days of the first dose of Modi-1ev/Modi-1eKv are eligible.
     * patient has refused SOC therapy (Modi-1ev/Modi-1eKv monotherapy cohort only).
   * SCCHN:

     o neoadjuvant expansion cohort only; patients who are treatment-naïve and are scheduled to have tumour resection surgery, in whom minimum of 3 weeks of Modi-1ev/Modi-1eKv and a single 400 mg intravenous (i.v.) total dose of pembrolizumab immunotherapy can be administered. Patients will only be enrolled once the Modi-1 Moditope® expansion doses and a lack of increased anti-CCP antibodies (with, and without, concomitant pembrolizumab) have been established.
   * HGSOC including fallopian tube and primary peritoneal cancers:

     * patient must be considered unsuitable for platinum chemotherapy, defined as recurrence/progression within 6 months of prior platinum-containing chemotherapy or patients in whom platinum therapy is no longer thought appropriate. Patient must have received no more than two non-platinum regimens, from the time the patient is considered unsuitable for platinum chemotherapy (Modi-1ev/Modi-1eKv monotherapy cohort only).
     * patient completing a course of systemic therapy for whom a subsequent SOC therapy is not yet indicated or appropriate and with measurable disease in accordance with RECIST 1.1 (Modi-1ev/Modi-1eKv monotherapy cohort only).
     * patient has refused SOC therapy (Modi-1ev/Modi-1eKv monotherapy cohort only).
   * RCC:

     * patient is untreated for advanced RCC (Modi-1ev/Modi-1eKv + CPI doublet cohort only).
     * patient has received first-line treatment consisting of anti-angiogenic therapy (Modi-1ev/Modi-1eKv monotherapy cohort).
     * patient has favourable or intermediate International Metastatic Renal-Cell Carcinoma Database Consortium (IMDC) risk score (Heng et al. 2013) (Modi-1ev/Modi-1eKv monotherapy cohort).
     * patient has intermediate or poor International Metastatic Renal-Cell Carcinoma Database Consortium (IMDC) risk score (Heng et al. 2013) and is eligible for SOC nivolumab with ipilimumab immunotherapy (Modi-1ev/Modi-1eKv + CPI doublet cohort only).
     * patient has stopped immunotherapy due to toxicity and with residual disease as measurable by RECIST 1.1 (Modi-1ev/Modi-1eKv monotherapy cohort only).
     * patient completing immunotherapy, for whom a subsequent SOC therapy is not yet indicated or appropriate and with measurable disease in accordance with RECIST 1.1 (Modi-1ev/Modi-1eKv monotherapy cohort only).
     * patient on active surveillance (Modi-1ev/Modi-1eKv monotherapy cohort only).
     * patient is eligible for SOC nivolumab with ipilimumab immunotherapy (Modi-1ev/Modi-1eKv + CPI doublet cohort only).
     * patient has refused SOC therapy (Modi-1ev/Modi-1eKv monotherapy cohort only).
3. Where applicable, patient has completed last dose of prior cancer therapy at least 4 weeks before the first dose of study treatment.
4. Patient has been fully vaccinated against COVID-19, the last vaccination being at least 14 days prior to the patient's first dose of IMP, except for those who have declined or are not eligible for COVID-19 vaccination.
5. Patient has recovered to Grade ≤1 (CTCAE v5.0) from the effects (excluding alopecia) of any prior therapy for their malignancies.
6. Patient has at least one measurable lesion per RECIST 1.1 criteria by computed tomography (CT) scan or magnetic resonance imaging (MRI) (non-neoadjuvant cohorts).
7. Wherever possible, patients not scheduled for curative intent resection surgery should have a fresh tumour biopsy (or have an archival biopsy [obtained within the past 5 years] if obtaining a fresh biopsy is not feasible) at baseline for molecular studies, and agree to a post-treatment biopsy (at Week 25 or one of the EOT visits), if feasible. Patients in the SCCHN neoadjuvant cohort must have both a fresh pre-treatment biopsy and agree to have their resected tumour analysed.
8. Patient is male or female and at least 18 years of age.
9. Patient has a life expectancy of more than 6 months.
10. Patient has an ECOG performance status of 0 or 1.
11. Patient has adequate organ function as determined by the following laboratory values: absolute neutrophil count ≥1.5 x 109/L, platelets ≥100 x 109/L, haemoglobin >90 g/L (>5.6 mmol/L), lymphocytes ≥ 1 x 109/L, serum creatinine ≤1.5 x upper limit of the normal range (ULN), serum total bilirubin ≤1.5 x ULN, serum transaminases (aspartate aminotransferase [AST]/alanine aminotransferase [ALT]) ≤2.5 x ULN or ≤5.0 x ULN if liver metastases present.
12. Patient must be able and willing to provide written informed consent prior to any study related procedure. (In the event that the patient is re-screened for study participation or if a protocol amendment alters the care of an ongoing patient, a new informed consent form must be signed).
13. Women of child-bearing potential must have a negative serum pregnancy test during Screening (and a urine test within the 7 days prior to Day 1) and be neither breastfeeding nor intending to become pregnant during study participation. Women of child-bearing potential must agree to use highly effective contraceptive methods prior to study entry, for the duration of study participation, and for 120 days after discontinuation of vaccine monotherapy or 5 months after use with a CPI (or longer if the Summary of Product Characteristics [SmPC] of the CPI requires it).
14. Men who are potentially fertile with partners of child-bearing potential must agree to use highly effective contraceptive methods for the duration of study participation, and for 120 days after discontinuation of vaccine monotherapy or 5 months after use with a CPI (or longer if the SmPC of the CPI requires it).
15. Patient must be willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.
16. Patient scheduled to receive a CPI (e.g., pembrolizumab alone or nivolumab alone or where applicable with ipilimumab) together with Modi-1ev/Modi-1eKv must have been clinically evaluated, have not received prior CPI therapy, and the CPI must be deemed an appropriate treatment for their disease according to the CPI's SmPC (this does not apply to the neoadjuvant SCCHN cohort).

EXCLUSION CRITERIA

1. Patient has symptomatic central nervous system metastases or carcinomatous meningitis.
2. Patient is taking any systemic steroid therapy (exceeding 10 mg/day of prednisolone or equivalent) or is on any other form of immune suppressant medication within 2 weeks prior to the first dose of IMP. Physiological doses of systemic steroids such as those for the management of adrenal insufficiency, topical and inhaled steroids, such as those for the management of asthma, and patients with hypothyroidism stable on hormone replacement, are permitted.
3. Patient has a history of malignancy other than the disease under study within 2 years prior to Screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 2-year overall survival rate >90%), such as adequately treated carcinoma-in-situ of the breast or the cervix, melanoma-in-situ, non-melanoma skin carcinoma, superficial bladder cancer, prostate cancer with Gleason grade ≤6 and prostate specific antigen within normal range or stage I endometrial cancer.
4. Patient is pregnant, lactating, or is expecting to conceive/father children within the duration of the study.
5. Patient has a concurrent illness which would preclude study conduct and assessment, including, but not limited to, uncontrolled medical conditions, uncontrolled and active infection (considered opportunistic, life threatening, or clinically significant), uncontrolled risk of bleeding, uncontrolled diabetes mellitus, pulmonary disease (including obstructive pulmonary disease and pulmonary fibrosis), alcoholic liver disease, or primary biliary cirrhosis.
6. Patient has New York Heart Association (NYHA) class III or IV heart disease, myocardial infarction or stroke within previous 6 months, a history of significant cardiac abnormality and/or significant abnormal baseline ECG readout, active ischaemia, or any other uncontrolled cardiac condition such as angina pectoris, clinically significant arrhythmia requiring therapy, uncontrolled hypertension, significant cerebrovascular disease, or congestive heart failure.
7. Patient has anti-CCP antibody levels classified as equivocal or positive according to NHS guidelines, i.e., ≥ the ULN, or has an active autoimmune disease that may impact on the study treatment in the opinion of the Investigator.
8. Patient has received a live vaccine within 28 days, or an influenza vaccine within 14 days prior to the first dose of IMP. The timing of any other vaccines should be assessed on a case-by-case basis by the Investigator prior to study enrolment.
9. Patient has a known history of human immunodeficiency virus (HIV), hepatitis B virus (HBV; surface antigen reactive) or hepatitis C (HCV; RNA detected).
10. COVID-19 vaccination within 14 days prior to the first dose of IMP.
11. Patient has a known current or recent history (within the last year) of substance abuse including illicit drugs or alcohol.
12. History of any of the following: drug-induced severe cutaneous adverse reaction (SCAR; including, but not limited to Stevens-Johnson syndrome/toxic epidermal necrolysis [SJS/TEN], or drug reaction with eosinophilia and systemic symptoms [DRESS]), or dose-limiting immune-mediated reactions (Modi-1ev/Modi-1eKv + CPI RCC cohort only).
13. Patient has a known hypersensitivity to the IMP under study or their excipients. Where SOC CPIs are planned to be given with the IMP, the patient must not have a known hypersensitivity to the CPIs or their excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2022-04-07 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of clinical and laboratory adverse events (AEs) | For the duration of the study (12 weeks after the final dose of study treatment)
  To measure the incidence of AEs of Modi-1 Moditope (as monotherapy and in combination with a CPI (e.g., pembrolizumab or nivolumab provided as standard of care) when administered intradermally
Cellular immune response to Modi-1 Moditope on IFNγ ELISpot assay | For the duration of the study (12 weeks after the final dose of study treatment)
  (i) the mean peptide-specific ELISpot response minus two standard deviations is greater than the mean pre-treatment peptide-specific response plus one standard deviation (of this mean); and (ii) the ELISpot response is more than 50 spots per million peripheral blood mononuclear cells.

SECONDARY OUTCOMES:
Imaging Response using RECIST 1.1 and iRECIST to Modi-1 Moditope in the non-neoadjuvant setting | For the duration of the study (12 weeks after the final dose of study treatment)
  To measure imaging response of Modi-1 Moditope in non-neoadjuvant cohorts, as monotherapy in patients with TNBC, advanced/unresectable HPV-negative SCCHN, HGSOC, or RCC and in combination with CPI therapy (e.g., pembrolizumab, nivolumab, Ipilimumab)
Overall survival | For the duration of the study (12 weeks after the final dose of study treatment)
  The overall survival will measured in patients vaccinated with Modi-1 Moditope either as monotherapy or in combination with checkpoint inhibitors in the target population.
Progression-free survival in patients vaccinated with Modi-1 Moditope | For the duration of the study (12 weeks after the final dose of study treatment)
  The progression-free survival will measured in patients vaccinated with Modi-1 Moditope either as monotherapy or in combination with checkpoint inhibitors in the target population.
Pathological response in the neoadjuvant setting in patients vaccinated with Modi-1 Moditope or Modi-1 Moditope + Pembrolizumab | For the duration of the study (6 weeks after resection surgery)
  Pathological response will be measured in tumour tissue of patients vaccinated with Modi-1 Moditope monotherapy or Modi-1 Moditope + Pembrolizumab in patients with SCCHN undergoing planned resection
Celluar immune response in the neoadjuvant setting in patients vaccinated with Modi-1 Moditope or Modi-1 Moditope + Pembrolizumab | For the duration of the study (6 weeks after resection surgery)
  Immune cells will be profiled and measured in tumour tissue of patients vaccinated with Modi-1 Moditope monotherapy or Modi-1 Moditope + Pembrolizumab in patients with SCCHN undergoing planned resection

OTHER OUTCOMES:
Immune cell profiling in tumour samples | For the duration of the study (12 weeks after the final dose of study treatment)
  Immune cells will be profiled from available biopsy tissue
Measurement of circulating tumour deoxyribonucleic acid (ctDNA) | For the duration of the study (12 weeks after the final dose of study treatment)
  ctDNA will be measured in blood in patients vaccinated with Modi-1 Moditope either as monotherapy or in combination with checkpoint inhibitors in the target population.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Ottensmeier, MD, Principal Investigator — The Clatterbridge Cancer Centre NHS Foundation Trust, United Kingdom
Locations (16):
- United Kingdom (16):
  - Brighton and Sussex University Hospital, Brighton, Default
  - Velindre Cancer Centre, Cardiff, Default
  - Edinburgh Cancer Centre (NHS Lothian), Edinburgh, Default
  - Royal Surrey NHS Foundation, Guildford, Default
  - Imperial College Healthcare NHS Trust, London, Default
  - Mount Vernon, London, Default
  - University College London Hospital NHS Foundation Trust, London, Default
  - Christie NHS Foundation Trust, Manchester, Default
  - Nottingham University Hospitals Cancer Centre, Nottingham, Default
  - Lancashire Teaching Hospitals NHS Foundation Trust, Preston, Default
  - Sheffield Teaching Hospital NHS Foundation Trust, Sheffield, Default
  - The Royal Marsden NHS Foundation Trust, Sutton, Default
  - Belfast City Hospital, Belfast
  - Addenbrooke's Hospital, Cambridge University Hospitals, Cambridge
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Liverpool
  - Torbay and South Devon NHS Foundation Trust, Torquay

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual patient data available